CLINICAL TRIAL: NCT02718365
Title: A Multi-center, Prospective, Randomized Controlled Clinical Trial: Comparison Between Wedge Resection and Segmentectomy in the Surgical Treatment of Ground Glass Opacity-dominant Stage IA Non-small Cell Lung Cancer
Brief Title: Comparison Between Wedge Resection and Segmentectomy for Ground Glass Opacity- Dominant Stage IA NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lunxu Liu, Professor and Chair of Department of Thoracic Surgery, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSCI002
Record Dates: First submitted 2015-10-04; First posted 2016-03-24 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Lung Neoplasms; Surgery
Keywords: Lung Neoplasms; Surgery; VATS; GGO; GGN; Segmentectomy; Wedge Resection; Prognosis
MeSH Terms: conditions — Lung Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Wedge resection
  Interventions: Procedure: Wedge resection
- Group B (Active Comparator): Segmentectomy
  Interventions: Procedure: Segmentectomy

INTERVENTIONS:
Procedure: Wedge resection — A wedge resection is the surgical removal of the lung tumor with a small portion of the lung that surrounds the tumor. Hilar and mediastinal lymph nodes should be resected or sampled.
  Arms: Group A
Procedure: Segmentectomy — A segmentectomy removes a segment of a lung lobe anatomically, or inclusion of a portion of adjacent segment, but does not remove the whole lung lobe. Hilar and mediastinal lymph nodes should be resected or sampled.
  Arms: Group B

SUMMARY:
The purpose of this study is to evaluate whether the long-term outcome and safety of wedge resection are comparable to segmentectomy for the surgical treatment of early stage (IA) non-small cell lung cancer (NSCLC). Zhang et al. performed a meta-analysis of 53 studies and suggested that sublobectomy achieved a survival rate comparable to lobectomy in a selected population of patients with Stage I NSCLC. However, one critical question needs to be addressed, that is, does sublobectomy require segmentectomy or wedge resection? Cho et al. reported that, for pulmonary ground glass opacity (GGO) nodules (Stage IA NSCLC), wedge resection achieved a 5-year survival rate of 98.6% in the pure GGO group and 95.5% in the mixed GGO group. Cho et al. cautioned against performing wedge resection for mixed GGO nodules with GGO component ≤ 75%, due to the high recurrence rate. When radiology shows that the GGO component is ≥75%, pathology usually finds that the lesions are non-invasive. Therefore, these lesions are potential candidates for wedge resection. This randomized clinical trial is to assess whether wedge resection can be established as a standard treatment for Stage IA NSCLC with tumor size ≤ 2 cm and GGO component ≥ 75%.

DETAILED DESCRIPTION:
1. Selection procedures: When a case meets the inclusion criteria and does not meet exclusion criteria, the research assistant of each research participating center will fill out the Eligibility Application Form and submit it to the Research Committee for reviewing whether the case is eligible for the trial. The following rules will be strictly applied:

   1. The application and confirmation of eligibility should be preoperatively completed and any postoperative application will not be accepted.
   2. If the Eligibility Application Form is incomplete, it must be returned to be completed; otherwise, it will not be accepted.
   3. After being approved by the Research Committee, the case will be assigned a number (Baseline Number, BN) and an Eligibility Confirmation Notice will be sent to the applicant.
   4. After each research participating center receives the Eligibility Confirmation Notice, the research assistant of each center is responsible for the custody and documentation.
   5. Once being selected for registration, the content of the Eligibility Application Form will be input into the database and the case's eligibility is not allowed to be cancelled, that is, the relevant information cannot be deleted from the database, unless the patient declines the information to be used in this study.
   6. The data center will not accept any duplicated applications for any single case. If this happens, the first registered data will be used (i.e., the first time BN).
   7. In cases of duplicated applications or registration errors, the research assistant of each research participating center shall contact the Research Committee as soon as possible for liaison and documentation.
2. Qualification of the responsible surgeons who participate in this study: the responsible surgeons who participate in this study shall meet the following qualifications: 1) at least have completed 20 cases of VATS segmentectomy; and 2) have passed the blind review of his/her video records of the surgery.
3. Criteria for confirming operation quality: for the case to be included in the analysis, the responsible surgeon shall submit the video or photo recordings of the surgery to the Research Committee for evaluation of the surgical procedures.
4. Rules for handling the excluded patients identified intraoperatively: if the responsible surgeon finds that the patient in operation meets the exclusion criteria, the case will be excluded and the surgeon will follow the routine clinical practice of the research participating center to decide subsequent treatments that are not specified in this study protocol.

ELIGIBILITY:
Inclusion criteria:

1. Preoperative thin-section computed tomography (TSCT) will fulfill all of the following conditions:

   * Lung cancer is suspected.
   * Lesion size is more than 5 mm but equal to or less than 20 mm.
   * Consolidation/tumor (C/T) ratio is equal to or less than 0.25.
   * The center of the tumor is located in the outer third of the lung field.
   * Preoperative TSCT estimates a surgical margin of more than1.5 cm or the tumor's diameter.
2. Preoperative clinical staging: T1a-T1bN0M0 (according to UICC2017-8thTNM staging).
3. R0 resectable in segmentectomy and wedge resections plus mediastinal lymph node resection.
4. Aged 18 to 75 years old.
5. No prior chemotherapy or thoracic radiation therapy for any malignant diseases.
6. Preoperative FEV1.0>=1.0 L.
7. Performance status of ECOG 0 or 1.
8. Preoperative ASA scoring (American society of anesthesiology) class I -III.
9. Sufficient organ functions.
10. The patient agrees to participate in the trial and signs the informed consent form.

Exclusion criteria:

1. Quit smoking <2 weeks.
2. Preoperative FEV1 < 50% of the expected value.
3. Mediastinal lymph node metastasis confirmed by biopsy.
4. Pregnant or lactating women.
5. Serious mental illness.
6. With other malignant disease history within 5 years.
7. With the history of unstable angina or myocardial infarction within 6 months.
8. With the history of cerebral infarction or cerebral hemorrhage within 6 months.
9. With the history of sustained systemic corticosteroid therapy within 1 month.
10. The patient requires simultaneous surgical treatment of other diseases.
11. TSCT shows that the lesion is located in the right middle lobe.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1382 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
5-year Progression-Free-Survival | From date of the recruitment, assessed up to 60 months

SECONDARY OUTCOMES:
3-year Progression-Free-Survival | From date of the recruitment, assessed up to 36 months
5-year overall survival | From date of the recruitment, assessed up to 60 months
Pulmonary function in the first year after surgery | From date of the 1 month\ 3 months\ 6 months\ 12 months after surgery in every recruited patient
30-day Morbidity and mortality rates | From date of the recruitment, assessed up to 30 days
10-year overall survival | From date of the recruitment, assessed up to 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Lunxu Liu, M.D., Ph.D., Principal Investigator — Department of Thoracic Surgery, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Zhang Y, Sun Y, Wang R, Ye T, Zhang Y, Chen H. Meta-analysis of lobectomy, segmentectomy, and wedge resection for stage I non-small cell lung cancer. J Surg Oncol. 2015 Mar;111(3):334-40. doi: 10.1002/jso.23800. Epub 2014 Oct 16. PMID 25322915
- [Background] Hida Y, Teramura K, Muto J, Ohtaka K, Hase R, Nakada R, Watanabe Y, Matsui Y, Kaga K. [Indication of limited pulmonary resection for small-sized lung cancer based on preoperative clinical data]. Kyobu Geka. 2012 Jan;65(1):52-7. Japanese. PMID 22314158
- [Background] Tsutani Y, Miyata Y, Nakayama H, Okumura S, Adachi S, Yoshimura M, Okada M. Appropriate sublobar resection choice for ground glass opacity-dominant clinical stage IA lung adenocarcinoma: wedge resection or segmentectomy. Chest. 2014 Jan;145(1):66-71. doi: 10.1378/chest.13-1094. PMID 24551879
- [Background] Cho JH, Choi YS, Kim J, Kim HK, Zo JI, Shim YM. Long-term outcomes of wedge resection for pulmonary ground-glass opacity nodules. Ann Thorac Surg. 2015 Jan;99(1):218-22. doi: 10.1016/j.athoracsur.2014.07.068. Epub 2014 Nov 15. PMID 25440277